CLINICAL TRIAL: NCT00209846
Title: A Prospective Randomised Double-Blind Parallel-Group Placebo-Controlled Study of Gaboxadol in Primary Insomnia
Brief Title: A Study of Gaboxadol in Primary Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10402
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-03-30 (Estimated); Status verified 2007-03

CONDITIONS: Primary Insomnia
Keywords: Primary insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gaboxadol

SUMMARY:
To evaluate the safety and tolerability of gaboxadol in primary insomnia.

DETAILED DESCRIPTION:
To obtain long-term safety data in elderly patients with gaboxadol.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of primary insomnia

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320
Dates: Start 2004-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Safety
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Please contact: Annelies van der Hammen Legters, Study Director — H. Lundbeck A/S
Locations (1):
- Non-US study, principal location:, Gothenburg, Sweden